CLINICAL TRIAL: NCT05321992
Title: Evaluating a Community-Based Behaviour Change Communication Model to Prevent Cholangiocarcinoma in Khon Kaen, Thailand
Acronym: eCHEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Khon Kaen University (Other); Global Alliance for Chronic Diseases (GACD) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0609004105; 13955 (Other: HiREB)
Record Dates: First submitted 2022-03-08; First posted 2022-04-11 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cholangiocarcinoma; Liver Fluke-Related Cholangiocarcinoma; Opisthorchiasis
Keywords: health education; community-based education; complex intervention
MeSH Terms: conditions — Cholangiocarcinoma; Opisthorchiasis; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Community (No Intervention): Participants in this arm will not be given the eCHEC program
- eCHEC Community (Active Comparator): Participants in this arm will be given the eCHEC program as their intervention
  Interventions: Behavioral: eCHEC program

INTERVENTIONS:
Behavioral: eCHEC program — The eCHEC program is the enhanced Community-based Health Education and Communication (CHEC) model to prevent O. viverrini in an effort to decrease cholangiocarcinoma (CCA) in Khon Kaen, Thailand
  Arms: eCHEC Community

SUMMARY:
Liver cancer, specifically cholangiocarcinoma (CCA), is very common in different areas in Thailand. Many factors make this cancer more common, such as liver fluke infection, older age, eating raw fish, family history of cancer, alcohol intake, taking certain medicines (praziquantel), low intake of fresh vegetable, and low education. In 2015, researchers from Khon Kaen University developed the Community-based Health Education and Communication (CHEC) program to prevent liver cancer caused by liver flukes in communities of the Khon Kaen province, Thailand.

The main aim of this 5-year research study is to enhance the CHEC program to prevent liver cancer, and test if it is effective in improving the knowledge and behaviours of community residents regarding how to prevent liver cancer. This study will take place in Khon Kaen, Thailand. Other aims are to:

1. Increase understanding in the community that make it difficult to prevent liver cancer, as well as community characteristics that can help prevent liver cancer;
2. Incorporate the program we develop in healthcare to prevent liver cancer in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* any individual residing in one of the 16 villages selected in the Khon Kaen province of Thailand, aged 20 and older

Exclusion Criteria:

* any individual 19 years or younger
* any individual not residing in one of the 16 pre-selected villages in the Khon Kaen province of Thailand

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Intake of raw fish | 12 months
  Mean difference in the self-reported frequency of intake of raw fish in the intervention group compared to the control group. Self reported, pre- and post- intervention.
Intake of fruits and vegetables | 12 months
  Mean difference in the self-reported frequency of intake of fruits and vegetables in the intervention group compared to the control group. Self reported, pre- and post- intervention.
Smoking | 12 months
  Difference in the proportion of smoking habits in the intervention group compared to the control group. Self reported, pre- and post- intervention.
Alcoholic beverage intake | 12 months
  Mean difference in the intake of alcoholic beverages in the intervention group compared to the control group. Self reported, pre- and post- intervention.
Praziquantel use | 12 months
  Difference in the proportion of use of the medication praziquantel (prescribed or self-medicated) in the intervention group compared to the control group. Self reported, pre- and post- intervention.
Stool test (proportion of stool test concentration) | 12 months
  Difference in the proportion of positive stool test of concentration of O. viverrini, pre- and post-intervention.
Stool test (mean concentration) | 12 months
  Difference in the mean concentration of O. viverrini in the stool test, pre- and post-intervention.
Stages of change for risk behaviours affecting the development of CCA. | 12 months
  Mean difference in the stages of change for risk behaviours in the intervention group compared to the control group. Self reported, pre- and post- intervention.

SECONDARY OUTCOMES:
Knowledge of preventative measures against CCA | 12 months
  Mean difference in knowledge score about in knowledge of preventative measures against CCA in the intervention group compared to the control group. Measured in questions included in the community survey.
BMI | 12 months
  Cardiobolic measure linked to developing cancer. Change in the mean body mass index calculated from height and weight (self-reported).
Waist circumference | 12 months
  Cardiobolic measure linked to developing cancer. Change in the mean waist circumference (measured with measuring tape)
Blood pressure | 12 months
  Cardiobolic measure linked to developing cancer. Change in the mean measured blood pressure (automated, validated device)
Health literacy | 12 months
  Mean difference in health literacy knowledge score in the intervention group compared to the control group. Self reported, pre- and post- intervention
Quality of life | 12 months
  Mean difference in quality of life in the intervention group compared to the control group. Self reported, pre- and post- intervention. Using the EuroQol-5 dimension-5 level (EQ-5D-5L) tool

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, MBBS, PhD, Principal Investigator — McMaster University; Pattapong Kessomboon, MD, PhD, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Phu Wiang, Changwat Khon Kaen, Thailand